CLINICAL TRIAL: NCT05126095
Title: Monitoring Skeletal Muscle Mass Using Cone-Beam Computed Tomography in Patients With Head and Neck Cancer Undergoing Chemoradiotherapy: Single-center Prospective Study
Brief Title: Monitoring Skeletal Muscle Mass Using CBCT in Patients With H&N Cancer Undergoing Chemoradiotherapy
Acronym: MELINOE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, YI PAN, Prof., Guangdong Provincial People's Hospital
Other Study IDs: KY-Q-2021-213
Record Dates: First submitted 2021-11-07; First posted 2021-11-18 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Head and Neck Cancer; Radiotherapy; Adverse Effect
Keywords: Cone-beam Computerized tomography; Skeletal Muscle Mass; Body weight; Malnutrition
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries; Body Weight; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trial cohort: CBCT: before radiotherapy and once a week during radiotherapy
  Body weight: before radiotherapy and once a week during radiotherapy
  The Patient-Generated Subjective Global Assessment (PG-SGA): before radiotherapy, 1st week, 3rd week and the last week during radiotherapy.
  Interventions: Radiation: Radical radiotherapy

INTERVENTIONS:
Radiation: Radical radiotherapy — Intensity-modulated radiation therapy (IMRT)

SUMMARY:
Chemoradiotherapy is the standard treatment for unresectable locally advanced head and neck cancer (HNC). However, malnutrition is present in 44-88% HNC patients during chemoradiotherapy, which leads to loss of skeletal muscle mass (SMM) and poor clinical outcomes. Timely assessment of SMM and early intervention of malnutrition are particularly important for HNC patients undergoing radiotherapy. However, body composition and skeletal muscle loss are not accurately reflected by the current assessment tools of malnutrition, which only measure body mass index and body weight loss.

Cone-beam CT (CBCT), a variation of traditional CT, is widely performed to ensure the appropriate position of the patients during radiotherapy. The previous study showed that measuring skeletal muscle areas and its changes using CBCT during radiotherapy is feasible. The hypothesis of this study is loss of SMM is associated with severe adverse effects in HNC patients during radiotherapy compared with body weight loss.

DETAILED DESCRIPTION:
This is a prospective observational phase II study. Patients with locally advanced HNC scheduled to receive radical radiotherapy are prospectively enrolled in this study. CBCT and body weight are obtained before radiotherapy and once a week during radiotherapy. Severe adverse effects including grade 3-4 mucositis, dermatitis, haematological toxicity, interruption of radiotherapy, delayed chemotherapy, and unplanned admission are recorded during radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HNC including Oral Cavity, Oropharyngeal, Nasopharynx, Hypopharyngeal, and Laryngeal Cancers
* Clinical stage II-IVa according to the American Joint Committee of Cancer (the seventh edition)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Exclusion Criteria:

* Previous head and neck radiotherapy
* Previous cervical lymph node dissection
* Active infections
* Palliative treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced HNC scheduled to receive radical radiotherapy
Sampling Method: Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-06-14 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
The treatment-related severe adverse events | 7 weeks
  The association between Loss of SMM and treatment-related severe adverse events including grade 3-4 mucositis, dermatitis, haematological toxicity, interruption of radiotherapy, delayed chemotherapy, and unplanned admission in HNC patients during radiotherapy.

SECONDARY OUTCOMES:
The weight loss percentage | 7 weeks
  The association between percentage Loss of SMM and weight loss percetage in HNC patients during radiotherapy
Scored Patient-Generated Subjective Global Assessment (PG-SGA) | 7 weeks
  The association between Loss of SMM and PG-SGA in HNC patients during radiotherapy. The PG-SGA scores typically range from 0-35, with a higher score reflecting a greater risk of malnutrition.
the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | 7 weeks
  The association between Loss of SMM and Quality Of Life in HNC patients during radiotherapy
the European Organization for Research and Treatment of Cancer Quality of Life Head and Neck Cancer Module (EORTC QLQ-H&N35) | 7 weeks
  The association between Loss of SMM and Quality Of Life in HNC patients during radiotherapy
Duration ofParenteral nutrition | 7 weeks
  The association between Loss of SMM and duration of parenteral nutrition in HNC patients during radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: YI PAN, Prof., Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- YI PAN, Guangzhou, Guangdong, China